CLINICAL TRIAL: NCT00660205
Title: Venous Thromboembolism and Haemostatic Disturbances in Patients With Upper Gastrointestinal Cancer
Acronym: GIVTE
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: N-20080002
Record Dates: First submitted 2008-04-10; First posted 2008-04-17 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Thrombosis; Deep Venous Thrombosis; Pulmonary Embolism; Venous Thromboembolism; Pancreas Cancer; Esophagus Cancer; Gastric Cancer
Keywords: DVT; PE; D-dimer; cancer; VTE
MeSH Terms: conditions — Thrombosis; Venous Thrombosis; Pulmonary Embolism; Venous Thromboembolism; Pancreatic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples with seperation in plasma and serum. Urin samples. tumour tissue samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- operation: Patients with upper gastro intestinal cancer who underwent surgery
- palliation: Patients with upper gastro intestinal cancer who did not underwent surgery
- control: Persons with no cancer who accepted to be control with blood samples and flow doppler ultrasound examination of both legs.

SUMMARY:
Cancer is a well known risk factor for venous thromboembolism (VTE) such as deep venous thrombosis (DVT) and pulmonary embolism (PE). Today we know that patients with adenocarcinomas of the gastro intestinal tract (GI-tract) often is in a hypercoagulable state.

In our observational study we collect patients admitted to department with a tentative diagnosis of upper GI cancer including pancreas cancer and offer them flow doppler ultrasounds of both legs for diagnosis of DVT in the entire treatment time. The routine CT-scan of the chest is modified to diagnose PE. This will be compared with blood samples analysed for coagulation markers including D-dimer - a fibrinogen degradation product.

DETAILED DESCRIPTION:
Armand Troussau observed back in 1865 a particular condition of the blood that predisposes to spontaneous coagulation in patients with gastric cancer. Today it is known that adenocarcinomas in the gastrointestinal (GI) tract including tumours of colon and rectum is accompanied by an hypercoagulable state.

Cancer is a well known risk factor for venous thromboembolism (VTE) such as deep venous thrombosis (DVT) and pulmonary embolism (PE). In fact PE in cancer patients is the second most common cause of death.

In an analysis of 13 cohort studies published with observational data Otten and Prins concludes that the prevalence of VTE in cancer patients varied between 10 and 20%. Variation could be explained with inconsistency. Patients suffering from thrombosis secondary to hemi paresis and paraplegia were included. Patients where included at time of VTE and not at time of cancer diagnosis.

Levitan et al looked at discharge diagnosis in 1211944 cancer patients and found among gastric cancer patients a frequency of VTE at 85 per 10000 patients and in pancreatic cancer 110 per 10000. Gastric cancer patients had a relative risk of 1.49 compared to non-cancer patients and pancreatic cancer patients a relative risk of 2.05 compared to non-cancer patients. This put pancreatic cancer among the most prone malignancy to cause thromboembolic complications. In a newly published study of 202 pancreatic cancer patients 19 developed venous thrombosis resulting in a 58 fold increased risk compared to general population with an incidence of 108/1000 patient-years and cumulative incidence after 6 months of 74/1000. 15 out of 19 cases of VTE occurred in the first 6 months since diagnosis of cancer. Tumours located in the corpus or cauda had twice the risk of caput. Chemotherapy resulted in a 4.8 fold risk of venous thrombosis.

Postoperatively VTE is higher in cancer patients than in non-cancer patients after surgery. A multicenter study including Danish patients - using phlebography - has shown VTE in 23% of patients after surgery for colorectal cancer. Coagulation activity - as assessed by sensitive biochemical markers - was related to tumour load.

Stender et al has in a newly published study shown a high preoperative prevalence of DVT in 193 colorectal cancer patients with a prevalence of 16% in women and 2.6% in men. In another newly published study asymptomatic DVT is found ovarian cancer patients with elevated levels of D-Dimer before treatment. The mechanism by which cancer induce VTE is at present subject to great interest.

Plasma D-dimer (DD), a degradation product of cross-linked fibrin, is routinely used to support or exclude the tentative diagnosis of DVT, combined with clinical assessment and ultrasonography (US).

The accuracy of DD assays in cancer patients is unknown, despite their high negative predictive values (NPV) in non cancer patients. A negative DD seems to exclude PE in cancer patients, but DD in combination imaging techniques such as US or computed tomography (CT) seems to improve diagnostic work-up but needs further investigation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of upper gastro intestinal cancer.

Exclusion Criteria:

* Earlier (within prev. 3 years) or concomitant cancer disease of any origin.
* Known immunological connective tissue disease.
* Mental disorder.
* Treatment with heparin, low molecular weight heparin or K-vitamin antagonist at the time of inclusion.
* Consent not attained.

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From February 2008 to December 2009 all patients admitted to The Department of Surgical Gastroenterology with upper GI cancer or pancreatic cancer will be included.
  Depending on the disease nature and progression, the patients will be followed as palliation or surgery cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2008-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ole Thorlacius-Ussing, Professor, DMSC, MD, Principal Investigator — Aalborg Hospital department of Aarhus University Hospital
Locations (1):
- Department of Surgical Gastroenterology, Aalborg Hospital, Aalborg, Region North, Denmark